CLINICAL TRIAL: NCT00600522
Title: Ultrasound-Guided Conservative Heopatecomy for Tumors Invading the Middle Hepatic Vein at the Caval Confluence as Alternative to Mesohepatectomy and Trisectionectomy
Brief Title: Alternative Surgical Policy for Central Liver Tumors
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Prof. Guido Torzilli, University of Milan - Istituto Clinico Humanitas, IRCCS
Other Study IDs: HEP-MHV; NEWHEP-2
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Colorectal Liver Metastases; Hepatocellular Carcinoma
Keywords: intraoperative ultrasonography; hepatectomy; colorectal liver metastases; hepatocellular carcinoma; contrast enhanced intraoperative ultrasonography.
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients selected for hepatectomy because carriers of hepatocellular carcinoma or colorectal cancer liver metastases invading the middle hepatic vein at caval confluence (last 4 cm).
  Interventions: Procedure: Ultrasound-guided hepatectomy

INTERVENTIONS:
Procedure: Ultrasound-guided hepatectomy — After laparotomy and staging by intraoperative ultrasound (IOUS), anterior surface of the hepatocaval confluence is exposed. Than, compression by means of the surgeon's finger-tip is applied at the MHV caval confluence verifying at color-Doppler IOUS the disappearance of the blood flow in the MHV or its inversion. Then, MHV clamping itself is carried out, and parenchymal sparing resection would be selected if at least one of these 3 findings is confirmed:
  1. Reversal color-Doppler IOUS flow direction in the peripheral portion of the MHV, which suggests the drainage through collateral circulation in the RHV/LHV depending on the side of the MHV branch with reversal flow.
  2. Detectable shunting collaterals at color-Doppler IOUS with RHV or LHV.
  3. Hepatopetal flow in P5-8 and/or P4inf portal branches. If none of these finding is confirmed and in particular hepatofugal flow direction in the P5-8 and/or P4 inf is detected the hepatectomy has to be extended.

SUMMARY:
Major hepatectomies have not negligible morbidity and mortality. However, when tumors invade middle hepatic vein (MHV) at caval confluence major surgery is usually recommended. Ultrasound-guided hepatectomy might allow conservative approaches. We prospectively check its feasibility in a series of patients carriers of tumors invading the MHV at the caval confluence.

DETAILED DESCRIPTION:
Major hepatectomies have not negligible morbidity and mortality. However, when tumors invade middle hepatic vein (MHV) at caval confluence trisectionectomy (TS) is generally performed, and central hepatectomy or mesohepatectomy (MH) (Segments 4, 5 and 8), is considered by some authors to be the conservative alternative to the previously cited approach. Between these two surgical interventions there is not, up to now, any evidence that one of them should be clearly preferred; anyway both are mojor resections. We previously reported that a surgical approach based on ultrasound-guided hepatectomy might minimize the need for major resection, whose rates of morbidity and mortality are not negligible. This policy could be useful also for disclosing new, more conservative, and better tolerated approaches for tumors invading the MHV at caval confluence in alternative to MH and TS. This study analyses the feasibility, safety and effectiveness of ultrasound-guided resections applied to these patients enrolled prospectively from a cohort of consecutive patients who undergo hepatectomy for tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients carriers of HCC or colorectal cancer liver metastases (CLM) who have macroscopic signs of vascular invasion (preoperative imaging and/IOUS) of the MHV close to the hepato-caval confluence (within 4 cm) demanding for that MHV resection.

Minimum follow-up for patients' inclusion was established at 6-months from surgery.

Exclusion Criteria:

* Patients carriers of tumors occupying entirely the right paramedian section and the segment 4, for whom at least a MH would have been compulsorily carried out.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients carriers of hepatocellular carcinoma or colorectal cancer liver metastases addressed to surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the rate of failure of conservative resection, i.e. the rate of patients who received TSs or MHs despite they fitted in the eligibility criteria. | January 2007

SECONDARY OUTCOMES:
The secondary outcome measure was the safety of the procedure. For that, we studied morbidity, mortality, amount of blood loss, rate of blood transfusions, and postoperative trend of liver function tests. | January 2007

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — University of Milan, Istituto Clinico Humanitas - IRCCS
Locations (1):
- Istituto Clinico Humanitas, IRCCS, Rozzano, Milano, Italy

REFERENCES:
- [Background] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Background] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Background] Stratopoulos C, Soonawalla Z, Brockmann J, Hoffmann K, Friend PJ. Central hepatectomy: the golden mean for treating central liver tumors? Surg Oncol. 2007 Aug;16(2):99-106. doi: 10.1016/j.suronc.2007.05.002. Epub 2007 Jun 20. PMID 17583496
- [Derived] Torzilli G, Palmisano A, Procopio F, Cimino M, Botea F, Donadon M, Del Fabbro D, Montorsi M. A new systematic small for size resection for liver tumors invading the middle hepatic vein at its caval confluence: mini-mesohepatectomy. Ann Surg. 2010 Jan;251(1):33-9. doi: 10.1097/SLA.0b013e3181b61db9. PMID 19858707